CLINICAL TRIAL: NCT02257268
Title: Effectiveness of VAMOS - a Change Behavior Program for Physical Activity and Healthy Eating Promotion - in Hypertensives
Brief Title: Effectiveness of a Program for Physical Activity and Healthy Eating Promotion in Hypertensives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Aline Mendes Gerage, PhD student, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAMOS REC 01
Record Dates: First submitted 2014-09-27; First posted 2014-10-06 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
Keywords: health behavior; risk factors;
MeSH Terms: conditions — Hypertension; Health Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Change behavior group (Experimental): Change behavior group = Group of change behavior including physical activity and healthy habits promotion.
  Interventions: Behavioral: VAMOS program - Active life improving health
- Control group (No Intervention): Control group = Group that will not receive the VAMOS program as intervention.

INTERVENTIONS:
Behavioral: VAMOS program - Active life improving health — All participants that will be assigned to change behavior group will participate of a change behavior program, entitled VAMOS (Active Life Improving Health), for 12 weeks. VAMOS is a lifestyle promotion program, that includes physical activity and healthy eating habits. The program is composed by a weekly meeting, in group, lasting about 90 min. In each weekly meeting, will be discussed guidelines and strategies for physical activities practices in different domains and for adoption of a healthy diet. All aspects and strategies included in the program are based in behavior changes theories. The participants of this group will receive an educational material and, in the middle of the program, they will earn a pedometer to aid in motivation and in the self-monitoring physical activity.
  Arms: Change behavior group

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of VAMOS program, a physical activity and healthy eating promotion program, in hypertensive from Recife-Pernambuco- Brazil. Approximately 90 subjects with a diagnosis of hypertension, under anti-hypertensive medication and classified as non-physically active, will be selected and randomly distributed into two groups: a change behavior group (CBG) and control group (CG). The CBG will participate of a change behavior program, entitled VAMOS - Active Life Improving Health, for 12 weeks and composed of a weekly meeting, in group, lasting about 90 minutes. In each weekly meeting, will be presented and discussed guidelines and strategies for practical physical activities in different fields and for adoption of a healthy diet in order that the level of physical activity and eating quality improve. The program will be evaluated by effectiveness, implementation and maintenance (initial and individual level) dimensions of RE-AIM framework. The effectiveness will be assessed from anthropometric measurements, body composition, eating habits, physical activity level, stages of self-change, self-efficacy, social support, quality of life and assessment of cardiovascular function at rest (clinic and home blood pressure, arterial stiffness, blood flow and flow-mediated dilation, heart rate and heart rate variability) before and after 12 weeks of intervention. The implementation will be assessed by identifying the extent to which the program will be conducted as planned. The maintenance, initial and at individual level, will be estimated from revaluations of all outcomes, as measured before and after the intervention, three months after the end of the program. For data analysis, in addition to descriptive statistics, two-way ANOVA for mixed models wil be applied for for within and between groups comparison, if the premises of this test are met. The level of significance that will be adopted is P<0.05. All analyzes will be done at SPSS statistical package, version 17.0.

DETAILED DESCRIPTION:
The overall goal of this study is to evaluate the effectiveness of VAMOS program, a physical activity and healthy eating promotion program, in hypertensive from Recife-PE- Brazil. As secondaries goals, the study attempts to:

1. evaluate the effectiveness of VAMOS program with regard to physical activity, the sedentary behavior and eating habits in hypertensives;
2. analyze whether self-efficacy, stages of self-change and social support mediate the possible effects of VAMOS program on physical activity, sedentary behavior and eating habits in hypertensives;
3. evaluate the effectiveness of VAMOS program with regard to clinic and home blood pressure, arterial stiffness, blood flow and flow-mediated dilation, heart rate and heart rate variability in hypertensives;
4. evaluate the effectiveness of VAMOS program on anthropometric and body composition variables in hypertensives;
5. analyze whether the possible result changes brought from VAMOS program in behavioral and biological variables promote changes in quality of life of hypertensives;
6. assess the implementation of VAMOS program in nonpharmacological treatment of hypertension in Recife, northeastern of Brazil;
7. identify whether the possible effects achieved from VAMOS remain three months after the end of the program in hypertensives.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension;
* Must be under anti-hypertensive medications for three months or more;
* May not present diabetes or other cardiovascular diseases;
* May not be engaged in regular physical activity;
* May not have physical disabilities that compromise the physical activity practices.

Exclusion Criteria:

* Not agree to participated with study;
* Not agree to sign the written informed consent;
* Change in doses or type of anti-hypertensive medications.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
change in clinic blood pressure | baseline, 12 weeks, 24 weeks
  Systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be checked using an automatic oscillometric instrument (Omron HEM 742-E0 - USA). The patients will be instructed to eat a light meal before the measurements, to avoid physical exercise and alcohol ingestion for at least 24 hours prior to the visit, and to avoid smoking and caffeine for at least 12 hours. Measurements will be taken in two non-consecutive days, after 10 minutes of rest in the supine position and three measurements will be done in each day, with one minute interval between measurements. All measurements will be taken on the left arm, in a quiet environment, with monitored temperature.
change in physical activity | baseline, 12 weeks, 24 weeks
  Habitual physical activity will be assessed by GT3X or GT3X+ accelerometer (Actigraph - USA) and Actilife 6.10 software will be used to analysis. Each participant will be instructed to use the accelerometer for seven consecutive days, removing it only for sleeping, bathing or performing water activities. The device will be attached to an elastic belt and fixed in the right side of the hip. Data will be collected in a 30 Hz sample frequency and will be analyzed using 60-s epochs. Periods with consecutive values of zero (with 2-min of spike tolerance) for 60 min or longer will be interpreted as "accelerometer not worn" and excluded from the analysis. Physical activity data only will be included if the participant accumulate a minimum of 10 hours/day of recording for at least four days, including one weekend day.
change in eating habits | baseline, 12 weeks, 24 weeks
  Eating habits will be investigated from the number of meals daily, quality chewing food, dietary intake concomitantly liquids at mealtimes, habit of eating salads, raw or cooked vegetables, daily water consumption habits and intake of visible fat from meat and chicken. Also, the food frequency questionnaire will be applied, using a list of foods for which the average frequency of consumption over the last three months is given.

SECONDARY OUTCOMES:
change in anthropometric parameters | baseline, 12 weeks, 24 weeks
  Body mass will be measured with participants wearing light clothes and no shoes, using an automatic scale (Welmy - Brazil) to the nearest 0.1 kg. Height will be measured using a stadiometer connected to scale to the nearest 0.5 cm. Body mass index will be calculated as the ratio between body mass in kilograms and the square of height in meters.
change in body composition | baseline, 12 weeks, 24 weeks
  Total body fat and body fat trunk will be estimated by densitometry scans for dual-energy X-ray absorptiometry (DXA) (Lunar Prodigy DXA, model NRL 41990, GE Lunar, Madison, WI). For the assessment, participants will be instructed to remain clothed but to remove any metallic prosthesis or objects. The procedure will last five to ten minutes for each individual and will be carried out by the same technician who will calibrate the device according to the manufacturer's recommendations.
change in arterial stiffness | baseline, 12 weeks, 24 weeks
  Pulse wave analyses, to obtain augmentation index, central systolic blood pressure, diastolic blood pressure and carotid-femoral pulse wave velocity will be measured using Sphygmocor (Atcor Medical, Sydney, Australia). The measurement of these parameters will be done according to guidelines specified by the Clinical Application of Arterial stiffness, Task Force III.
change in heart rate variability | baseline, 12 weeks, 24 weeks
  For heart rate variability assessment, R-R interval will be obtained using a heart rate monitor (POLAR, RS 800CX; Polar Electro Oy Inc, Kempele, Finland). Participants should remain in the supine position for 10 minutes, after approximately 10 minutes at rest. All analyses will be performed with Kubios software (Biosignal Analysis and Medical Imaging Group - Finland) by a single evaluator, following the recommendations of the Task Force of the European Society of Cardiology and the North American.
change in blood flow and flow-mediated dilation | baseline, 12 weeks, 24 weeks
  For assessment of blood flow and flow-mediated dilation, the method of venous occlusion pletysmography will be used (Hokanson - EC6 - EUA) with measurement being done in the left arm. A cuff will be placed around the left arm and another cuff will be placed around the wrist. A strain gauge pletysmography will be positioned in the largest forearm circumference. For blood flow measurement, the wrist cuff will be inflated and then the arm cuff for 10 seconds, followed by 10 seconds of deflation, totaling 20 seconds in each cycle. Inflation of the cuff will be made during the cardiac diastole, which will be perceived by an electrocardiogram. The measurement will be performed 12 times in a row, completing four minutes. The flow-mediated vasodilation will be assessed by vascular response to vasodilator stimuli using the technique of reactive hyperemia.
change in home blood pressure monitoring | baseline, 12 weeks, 24 weeks
  Each participant will receive an automatic device (OMRON - HEM - 742INT) and will be instructed to perform over four days, four measures of blood pressure at home, two in the morning and two at night. They will be instructed to taking five minutes of rest and one minute of interval between measurements. In addition, subjects will be instructed to perform the steps before taking the medicaments and before breakfast or dinner, following the recommendations of III Guidelines for Home Blood Pressure Monitoring.
change in stages of self-changes | baseline, 12 weeks, 24 weeks
  The stages of self-changes for physical activity and for healthy eating habits will be assessed by questionnaires that classified subjects in one of five stages: pre-contemplation, contemplation, preparation, action and maintenance.
change in self-efficacy | baseline, 12 weeks, 24 weeks
  The self-efficacy will be evaluated by scale "Self-Efficacy to Regulate Eating Habits e Self-Efficacy to Regulate Exercise" proposed by Bandura (2006) and validated for Brazilian adults by Boff (2012).
change in social support | baseline, 12 weeks, 24 weeks
  The social support for physical activities will be evaluated by a scale proposed by Reis et al. (2011).
change in quality of life | baseline, 12 weeks, 24 weeks
  The quality of life will be assessed by two general questions from Whoqol BREF.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael M Ritti-Dias, Doctor, Study Director — University of Pernambuco; Tania Rosane B Benedetti, Doctor, Study Director — Federal University of Santa Catarina; Aline M Gerage, PhD student, Principal Investigator — Federal University of Santa Catarina
Locations (1):
- Aline Mendes Gerage, Florianópolis, Santa Catarina, Brazil

REFERENCES:
- [Derived] Gerage AM, Benedetti TRB, Cavalcante BR, Farah BQ, Ritti-Dias RM. Efficacy of a behavior change program on cardiovascular parameters in patients with hypertension: a randomized controlled trial. Einstein (Sao Paulo). 2020 Jan 31;18:eAO5227. doi: 10.31744/einstein_journal/2020AO5227. eCollection 2020. PMID 32022106
- [Derived] Gerage AM, Benedetti TRB, Ritti-Dias RM, Dos Santos ACO, de Souza BCC, Almeida FA. Effectiveness of a Behavior Change Program on Physical Activity and Eating Habits in Patients With Hypertension: A Randomized Controlled Trial. J Phys Act Health. 2017 Dec 1;14(12):943-952. doi: 10.1123/jpah.2016-0268. Epub 2017 Sep 22. PMID 28682707